CLINICAL TRIAL: NCT05216640
Title: High Flow Nasal Cannula Versus High Velocity Nasal Insufflation in Covid-19 Patients Admitted to Respiratory Intensive Care Unit of Assiut University Hospital
Brief Title: High Flow Nasal Cannula Versus High Velocity Nasal Insufflation in Covid-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Basma Abd ElAziz Mohammed, Resident doctor, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HFNC VS HVNI in COVID 19
Record Dates: First submitted 2021-11-13; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; Acute Respiratory Failure
Keywords: HFNC; HVNI
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Nasal Cannula (Active Comparator): Standard operating procedures represented by high flow nasal cannula oxygen therapy
  Interventions: Device: High Flow Oxygen Therapy
- High Velocity Nasal Insufflation (Active Comparator): Standard operating procedures represented by high velocity nasal insufflation therapy
  Interventions: Device: High Flow Oxygen Therapy

INTERVENTIONS:
Device: High Flow Oxygen Therapy — • The patient will be allocated into 2 groups, patients who will require ventilatory support via HFNC and those who will require HVNI

SUMMARY:
To compare the outcomes of HFNC and HVNI in COVID-19 patients with acute respiratory failure as regard need for mechanical ventilation, changes of arterial blood gases (ABG) parameters, duration of ventilatory support and delay between admission and intubation

DETAILED DESCRIPTION:
novel clinical syndrome caused by a previously unknown coronavirus, SARS-Cov-2, was first identified in Wuhan (China) in December 2019. Despite massive efforts to contain viral transmission, a worldwide epidemic has developed from this virus. This disease is presently known as COVID-19 COVID-19 pandemic reached over 45 million confirmed infections and claimed the lives of more than 1.2 million people worldwide. The clinical features of COVID-19 are diverse and range from asymptomatic to critical illness and death. Severe and critical cases represented 14% and 5% of laboratory-confirmed COVID-19 patients and need ICU admission Several non-invasive options exist to support COVID-19 patients with mild or moderate respiratory distress and may reduce the numbers of patients requiring intubation, mechanical ventilation in some severely ill patients such as High flow nasal oxygen (HFNO) High flow nasal oxygen (HFNO) includes high flow nasal cannula and high velocity nasal insufflation. High flow oxygen systems provide oxygen-rich heated humidified gas to the patient's nose at flow levels sufficient to deliver a constant, precisely set high FiO2. Exhalation is to the open air. HFNO reduces dead space, provides low levels of PEEP, and decreases breathing frequency and work of breathing HFNC flow rates reach up to 60 L/min, whereas HVNI delivers flow rates up to 40 L/min due to differing mechanisms of delivery (4).

High velocity nasal insufflation (HVNI) utilizes a small-bore nasal cannula to generate higher velocities of gas delivery than HFNC which uses large bore cannula

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 positive by RT-PCR
* Age≥ 18 years
* Both gender
* Classical radiological lesions of COVID-19 on HRCT chest.
* Respiratory rate > 30/ min and not responding to non-rebreather masks.
* COVID-related pneumonia requiring non-invasive ventilatory support (high-flow nasal cannula, and / or non-invasive ventilation and / or CPAP)

Exclusion Criteria:

* Age < 18 years
* Patients who refuse to participate in the study
* Severe respiratory failure requiring invasive ventilatory support
* Indication of immediate tracheal intubation
* Significant acute progressive circulatory insufficiency
* Impaired conscious level
* Nasal blockade

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
To compare the outcomes of HFNC and HVNI in COVID-19 patients with acute respiratory failure | baseline
  need for mechanical ventilation
changes of arterial blood gases (ABG) parameters | within 2 hours then according to clinical condition
  changes of arterial blood gases (ABG) parameters
duration of ventilatory support | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  duration of ventilatory support
delay between admission and intubation. | baseline
  delay between admission and intubation.

SECONDARY OUTCOMES:
To evaluate the length of ICU stay and mortality rate in HFNC versus HVNI in COVID-19 patients | baseline
  duration of ICU stay
mortality rate | baseline
  mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Maha k Ghanem, MD, Study Director — Assuit university, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Wang Y, Chen Y, Qin Q. Unique epidemiological and clinical features of the emerging 2019 novel coronavirus pneumonia (COVID-19) implicate special control measures. J Med Virol. 2020 Jun;92(6):568-576. doi: 10.1002/jmv.25748. Epub 2020 Mar 29. PMID 32134116
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Alhazzani W, Moller MH, Arabi YM, Loeb M, Gong MN, Fan E, Oczkowski S, Levy MM, Derde L, Dzierba A, Du B, Aboodi M, Wunsch H, Cecconi M, Koh Y, Chertow DS, Maitland K, Alshamsi F, Belley-Cote E, Greco M, Laundy M, Morgan JS, Kesecioglu J, McGeer A, Mermel L, Mammen MJ, Alexander PE, Arrington A, Centofanti JE, Citerio G, Baw B, Memish ZA, Hammond N, Hayden FG, Evans L, Rhodes A. Surviving Sepsis Campaign: guidelines on the management of critically ill adults with Coronavirus Disease 2019 (COVID-19). Intensive Care Med. 2020 May;46(5):854-887. doi: 10.1007/s00134-020-06022-5. Epub 2020 Mar 28. PMID 32222812
- [Background] Nishimura M. High-Flow Nasal Cannula Oxygen Therapy in Adults: Physiological Benefits, Indication, Clinical Benefits, and Adverse Effects. Respir Care. 2016 Apr;61(4):529-41. doi: 10.4187/respcare.04577. PMID 27016353
- [Background] Doshi P, Whittle JS, Bublewicz M, Kearney J, Ashe T, Graham R, Salazar S, Ellis TW Jr, Maynard D, Dennis R, Tillotson A, Hill M, Granado M, Gordon N, Dunlap C, Spivey S, Miller TL. High-Velocity Nasal Insufflation in the Treatment of Respiratory Failure: A Randomized Clinical Trial. Ann Emerg Med. 2018 Jul;72(1):73-83.e5. doi: 10.1016/j.annemergmed.2017.12.006. Epub 2018 Jan 6. PMID 29310868